CLINICAL TRIAL: NCT07177027
Title: The Effects of Breathing Exercises and Music Intervention During Labor on Pain Perception, Birth Expectations, and Birth Satisfaction in Primiparous Women: A Randomized Controlled Trial
Brief Title: The Effects of Breathing Exercises and Music Intervention During Labor on Pain Perception, Birth Expectations, and Birth Satisfaction in Primiparous Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Şeyma Çatalgöl, Dr, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 480-480-27
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Music Intervention; Breathing Exercises
Keywords: Music intervention; Breathing exercises; Birth; Pregnancy
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music intervention group (Experimental): In the music intervention group, participants were introduced to 12 music tracks at 36 weeks of gestation during childbirth preparation classes. Short samples of these tracks were played during the class, and the full tracks were then shared with participants via WhatsApp to encourage regular listening at home.
  During the prenatal period, participants received regular WhatsApp reminders every few days to listen to the music.
  During labor, participants were encouraged to listen to music whenever they wished. Additionally, at 4 cm, 6 cm, and 8 cm cervical dilation, all participants in this group listened to their preferred tracks from the playlist for 20 minutes. Pain intensity was measured using the Visual Analog Scale (VAS) before and after each music session. In the postpartum period, the Birth Expectation Scale and Birth Satisfaction Scale were administered.
  Interventions: Behavioral: Music intervention
- Breathing Exercises Group (Experimental): In the breathing exercise group, Lamaze breathing techniques were taught during prenatal classes and practiced throughout the labor process. They were encouraged to practice these exercises throughout labor. At 4, 6, and 8 cm cervical dilation, guided breathing exercises were conducted, and pain was assessed using the Visual Analog Scale (VAS) before and after each exercise.
  Interventions: Behavioral: Breathing Exercise
- Control Group (No Intervention): In the control group, participants received routine maternity care. VAS pain assessments were conducted at the same cervical dilation points (4, 6, and 8 cm), without any additional interventions. In the postpartum period, the Birth Expectation Scale and Birth Satisfaction Scale were administered.

INTERVENTIONS:
Behavioral: Music intervention — Participants listened to 12 relaxing music tracks introduced during prenatal childbirth classes at 36 weeks of gestation. The tracks were shared via WhatsApp to encourage regular listening during pregnancy. During labor, participants were encouraged to listen to music whenever they wished. At cervical dilations of 4 cm, 6 cm, and 8 cm, participants listened to their preferred tracks from the playlist for 20 minutes. Pain intensity was measured before and after each session using the Visual Analog Scale (VAS).
  Arms: Music intervention group
Behavioral: Breathing Exercise — Participants were trained in Lamaze breathing techniques during prenatal childbirth classes. They practiced guided breathing exercises during labor at cervical dilation points of 4 cm, 6 cm, and 8 cm. Pain intensity was assessed before and after each session using the Visual Analog Scale (VAS).
  Arms: Breathing Exercises Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of music listening and breathing exercises during labor on pain perception, birth expectations, and birth satisfaction among primiparous women. This randomized controlled trial was conducted in the delivery unit of a hospital located in the Inner Aegean Region of Turkey. The study included 90 primiparous pregnant women admitted for vaginal delivery. Participants without visual, auditory, or neurological impairments were included and randomly assigned into three groups: music intervention group, breathing exercise group, and control group (n=30 in each group).

Participants were randomly assigned to one of three groups (Music Intervention, Breathing Exercise, Control) using a computer-generated randomization sequence. Allocation concealment was ensured by using sealed, opaque envelopes prepared by a researcher who was not involved in participant recruitment or assessment.

In the music intervention group, participants were introduced to 12 music tracks at 36 weeks of gestation during childbirth preparation classes. Short samples of these tracks were played during the class, and the full tracks were then shared with participants via WhatsApp to encourage regular listening at home.

During the prenatal period, participants received regular WhatsApp reminders every few days to listen to the music.

During labor, participants were encouraged to listen to music whenever they wished. Additionally, at 4 cm, 6 cm, and 8 cm cervical dilation, all participants in this group listened to their preferred tracks from the playlist for 20 minutes. Pain intensity was measured using the Visual Analog Scale (VAS) before and after each music session.

In the breathing exercise group, Lamaze breathing techniques were taught during prenatal classes and practiced throughout the labor process. They were encouraged to practice these exercises throughout labor. At 4, 6, and 8 cm cervical dilation, guided breathing exercises were conducted, and pain was assessed using the Visual Analog Scale (VAS) before and after each exercise.

In the control group, participants received routine maternity care. VAS pain assessments were conducted at the same cervical dilation points (4, 6, and 8 cm), without any additional interventions.

For all participants, the durations of the first, second, and third stages of labor were recorded and compared across groups. In the postpartum period, the Birth Expectation Scale and Birth Satisfaction Scale were administered.

Study data included sociodemographic information, VAS pain scores, and scores from the birth expectation and satisfaction scales.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effects of music listening and breathing exercises during labor on pain perception, birth expectations, and birth satisfaction among primiparous women. The study was conducted in the delivery unit of a hospital in the Inner Aegean Region of Turkey and included 90 healthy primiparous pregnant women admitted for vaginal delivery. Participants who met the inclusion criteria were randomly assigned to one of three groups: music intervention group, breathing exercise group, or control group, with 30 women in each group.

Participants were randomly assigned to one of three groups (Music Intervention, Breathing Exercise, Control) using a computer-generated randomization sequence. Allocation concealment was ensured by using sealed, opaque envelopes prepared by a researcher who was not involved in participant recruitment or assessment.

In the music intervention group, participants attended childbirth preparation classes at 36 weeks of gestation, where they were introduced to 12 carefully selected music tracks. In order to determine the music pieces to be used in the study, a playlist consisting of 36 tracks with varying tempos and emotional content was created. The playlist included an equal number of slow, moderate, and fast-tempo pieces, each further divided into subcategories representing calming, neutral, and uplifting emotional tones.

The selection process involved 20 volunteer pregnant individuals who were not part of the study sample but shared similar demographic characteristics. These volunteers were asked to listen to short excerpts (30-60 seconds) of each track and to identify the 12 pieces they liked the most. Preferences were recorded either through a Likert-type rating form.

To minimize order effects, the music tracks were presented in a randomized sequence. Participants were encouraged to use headphones to reduce environmental distractions and ensure consistent audio quality.

This participant-based music selection approach was designed to enhance emotional and cultural alignment between the selected music and the target population. It also aimed to increase the ecological validity of the intervention by incorporating music preferences that are more likely to elicit genuine emotional and physiological responses.Short samples of each track were played during the class. The full music playlist was shared with each participant via WhatsApp for home listening, and regular reminders were sent every few days to encourage consistent use during the antenatal period. During labor, women were encouraged to listen to music freely. In addition, at 4, 6, and 8 cm of cervical dilation, all participants in this group were asked to listen to their preferred tracks from the playlist for 20 minutes. Pain intensity was evaluated before and after each listening session using the Visual Analog Scale (VAS).

In the breathing exercise group, participants were trained in Lamaze breathing techniques during childbirth preparation classes and were encouraged to apply these techniques throughout labor. At 4, 6, and 8 cm cervical dilation, structured breathing exercises were performed, and pain was assessed before and after each session using the VAS.

The control group received routine maternity care without any additional non-pharmacological interventions. However, VAS pain assessments were still conducted at 4, 6, and 8 cm cervical dilation for comparison.

The duration of the first, second, and third stages of labor was recorded for all participants. In the postpartum period, the Birth Expectation Scale and Birth Satisfaction Scale were administered to assess maternal perspectives and satisfaction with the birth experience.

Study data were collected using a sociodemographic data form, VAS for pain assessment, and validated scales for measuring birth expectations and satisfaction. The results of this study may inform the use of non-pharmacological interventions to improve maternal comfort and the childbirth experience in clinical practice.

ELIGIBILITY:
Inclusion Criteria:Participants were included in the study if they met the following criteria:

Voluntary participation in the study and provision of written informed consent, Being a primiparous pregnant woman, Aged between 18 and 35 years, Gestational age between 38 and 42 weeks, Ability to read and write, No hearing impairment that would prevent listening to music, Planning to deliver vaginally, No respiratory disorders (e.g., asthma, COPD) that would interfere with breathing exercises, No obstetric complications that could affect labor progression (e.g., precipitous labor, prolonged labor), Attendance in antenatal childbirth education classes, including learning breathing exercises and listening to the music pieces planned for the intervention.

Not receiving any labor-inducing medications

-

Exclusion Criteria: Participants were excluded if they met any of the following:

Withdrawal of consent or unwillingness to continue cooperation at any stage of the study, Refusal to continue with breathing exercises or music intervention during any phase of labor, Undergoing cesarean section due to medical indications despite initial plan for vaginal delivery, Gestational age outside of 38-42 weeks, Development of labor-related complications such as precipitous or prolonged labor during the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity During Labor | At 4 cm, 6 cm, and 8 cm cervical dilation during active labor
  Measurement Tool: Visual Analog Scale (VAS), 0-10 Description: Pain intensity will be assessed before and after each intervention session (music or breathing exercises) at specified cervical dilations. In the control group, VAS will be measured at the same points without intervention.
  Primary Purpose: To determine the effect of music and breathing interventions on perceived pain intensity during labor.
Duration of Labor Stages | During the first, second, and third stages of labor
  The duration (in minutes) of each labor stage will be recorded and compared between the three groups (music, breathing, and control).

SECONDARY OUTCOMES:
Within 6-12 hours postpartum | Within 6-12 hours postpartum
  Measurement Tool: Birth Expectation Scale Evaluates whether the birth experience met the woman's expectations, measured after delivery.
Birth Satisfaction Score | Within 6-12 hours postpartum
  Measurement Tool: Birth Satisfaction Scale , assesses overall maternal satisfaction with the birth experience.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma ÇATALGÖL, Dr, Principal Investigator — Uşak University
Locations (1):
- Uşak University, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No